CLINICAL TRIAL: NCT04057469
Title: Effect of Tulobuterol Patch Versus Placebo on the Occurrence of Respiratory Adverse Events in Children Undergoing Tonsillectomies
Brief Title: Tulobuterol Patch in Pediatric Patients Undergoing Tonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medical Center (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Severance Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1905-178-103
Record Dates: First submitted 2019-08-12; First posted 2019-08-15 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Tonsillar Hypertrophy
MeSH Terms: interventions — tulobuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tulobuterol patch (Experimental)
  Interventions: Drug: Tulobuterol Hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo transdermal patch

INTERVENTIONS:
Drug: Tulobuterol Hydrochloride — The appropriate time interval between the patch attachment and the end of surgery was within 8 to 10 hours.
  Arms: Tulobuterol patch
Drug: Placebo transdermal patch — The appropriate time interval between the patch attachment and the end of surgery was within 8 to 10 hours.
  Arms: Placebo

SUMMARY:
* Tonsillectomy is a common pediatric procedure for the treatment of sleep-disordered breathing and chronic tonsillitis. Up to half of children having this procedure experience a perioperative respiratory adverse event.
* We tried to determine whether tulobuterol patch (transdermal bronchodilator) premedication decreases the risk of perioperative respiratory adverse events in children undergoing anesthesia for tonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing tonsillectomy

Exclusion Criteria:

* recent upper respiratory infection (2weeks)
* Allergy to tulobuterol patch
* Patients receiving catecholamine (epinephrine, isoproterenol)
* hyperthyroidism
* hypertension
* cardiac disease
* Diabetes melitus
* atopic dermatitis
* Asthma

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
perioperative respiratory complication | from anesthetic induction to postanesthesia care unit discharge, an average of 3 hours
  laryngospasm, bronchospasm, oxygen desaturation, airway obstruction, severe coughing, postoperative stridor

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Hyun-Joo Kim, Seoul
  - Jin-Kyung Kim, Seoul
  - Chung-Ang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim EH, Lee SH, Kim JK, Park YH, Kang P, Park JB, Ji SH, Jang YE, Lee JH, Kim JT, Kim HS. Effect of Tulobuterol Patch Versus Placebo on the Occurrence of Respiratory Adverse Events in Children Undergoing Tonsillectomies: A Randomized Controlled Trial. Anesth Analg. 2023 Jun 1;136(6):1067-1074. doi: 10.1213/ANE.0000000000006355. Epub 2023 May 19. PMID 36727868